CLINICAL TRIAL: NCT04301856
Title: Evaluation of the Response to CFTR Modulators in Patients With Cystic Fibrosis Less Than 18 Years of Age
Brief Title: Response to CFTR Modulators in CF Patients Under 18 Years
Acronym: MODUL-CF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Societe Francaise de la Mucoviscidose (Other)
Responsible Party: Principal Investigator, Isabelle SERMET-GAUDELUS, Professor Isabelle Sermet-Gaudelus, Societe Francaise de la Mucoviscidose
Other Study IDs: 0011928
Record Dates: First submitted 2020-02-21; First posted 2020-03-10 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Cystic Fibrosis in Children
MeSH Terms: interventions — lumacaftor, ivacaftor drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Excess bronchial secretions and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CF children treated with CFTR modul: Cystic fibrosis patients under 18 years treated with CFTR modulators according to french health recommendations observational cohort study
  Interventions: Drug: CFTR Modulators

INTERVENTIONS:
Drug: CFTR Modulators — CFTR modulators as recommended in routine care by the french health authorities
  Other Names: Orkambi, Kalydeko...

SUMMARY:
CFTR modulators should improve the prognosis of Cystic Fibrosis. Identifying patients under the age of 18 responding to CFTR modulators as well as detecting possible toxicity is an important medical objective given the potential side effects and the high cost of these molecules.

This observational follow-up cohort study is carried out as part of routine care.

The main objective is to assess the evolution of pulmonary structural impairment by low-dose CF scan at the end of the first year of CFTR modulator therapy.

The secondary objectives are to evaluate structural impairment at low dose scan at 3 years and 5 years of CFTR modulator treatment, the evolution of respiratory functional parameters, growth, puberty, lung infection, sweat test, quality of life and pancreatic function, as well as tolerance of modulators including liver toxicity.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is a deadly disease. This is due to overinfected chronic obstructive pulmonary disease that progresses to end-stage respiratory failure. CFTR modulators should improve the prognosis of CF, as they may slow the progression of patients' lung disease. Assessing their impact in the paediatric population is becoming a major issue. Children and adolescents under the age of 18 are a target cohort because they have a lung disease that is still poorly developed. Early prescription of CFTR modulators is therefore a priority but requires evidence of absence of toxicity. Identifying patients under the age of 18 responding to CFTR modulators as well as detecting possible toxicity, is an important medical objective given the potential side effects and the high cost of these molecules.

The outcomes previously used in Phase III studies (FEV1, frequency of exacerbations, nutritional status) are insufficiently sensitive in this population.

Other criteria need to be analyzed to identify the response to CFTR modulators in the short and medium term. The investigators hypothesize that the assessment of pulmonary structural impairment by low-dose lung CT-scan as part of routine care could be a much more sensitive criterion for the development of lung disease under CFTR modulators.

This observational follow-up cohort study is carried out as part of routine care. It does not involve a specific collection for research. Excess bronchial secretions and blood will be kept instead of being discarded in the event of a possible requalification for research.

The main objective is to assess the evolution of pulmonary structural impairment by low-dose CF scan at the end of the first year of CFTR modulator therapy The secondary objectives are to assess following criteria

* Tolerance of modulators in this age group, including screening for bronchial reactivity at treatment, early liver toxicity
* Longitudinal evolution of pulmonary structural impairment by low dose scan at 3 years and 5 years of CFTR modulator treatment
* Evolution of respiratory functional parameters
* Measurement by spirometry and plethysmography
* Lung clearance index (if possible)
* Longitudinal evolution of bacterial colonization, compared to the year prior to modulating treatment
* Exacerbations: number, duration, days of antibiotics, hospitalizations, return to stable condition
* Colonization of bronchial secretions
* Changes in quality of life
* Evolution of the sweat test
* Longitudinal evaluation of pancreatic function
* Longitudinal evaluation of growth and puberty compared to the year prior to CFTR modulator
* Growth speed, and bone age
* Bone mineralization, body composition (if possible)
* Pubertal markers from 9 years in girls and 10 years in boys
* Evaluation of glycemic dysregulation if present
* Preservation of samples taken as part of routine care (serum, bronchial secretions) for possible research use

ELIGIBILITY:
Inclusion Criteria:

Children with cystic fibrosis under the age of 18 under CFTR modulator therapy

Exclusion Criteria:

* Patients with cystic fibrosis without indication for CFTR modulator therapy
* Patients over the age of 18
* Pregnant or lactating women

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with cystic fibrosis under the age of 18 eligible for CFTR modulator thérapies according to french national recommandations
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Lung Imaging | at initiation, as part of national guidelines
  Lung structural injury assessed by Low Dose CT, as part of routine care
Lung Imaging | at 1 year, as part of national guidelines
  Lung structural injury assessed by Low Dose CT, as part of routine care
Lung Imaging | at 3 years, as part of national guidelines
  Lung structural injury assessed by Low Dose CT, as part of routine care
Lung Imaging | at 5 years, as part of national guidelines
  Lung structural injury assessed by Low Dose CT, as part of routine care

SECONDARY OUTCOMES:
weight in kilogrammes | longitudinal monitoring of assessments carried out as part of routine care during 5 yrs
  weight in kilogrammes (associated with a retrospective collection in the year prior to treatment)
height in meters | longitudinal monitoring of assessments carried out as part of routine care during 5 yrs
  height in meters (associated with a retrospective collection in the year prior to treatment)
pubertal evolution | longitudinal monitoring of assessments carried out as part of routine care during 5 yrs
  pubertal evolution (associated with a retrospective collection in the year prior to treatment)
bronchial infectious exacerbations | longitudinal monitoring of assessments carried out as part of routine care during 5 yrs
  bronchial infectious exacerbations (associated with a retrospective collection in the year prior to treatment)
Forced Expiratory Volume in 1 second(FEV1) | longitudinal monitoring of assessments carried out as part of routine care during 5 yrs
  Forced Expiratory Volume in 1 second(FEV1) in liter
Forced Vital Capacity (FVC) | longitudinal monitoring of assessments carried out as part of routine care during 5 yrs
  Forced Vital Capacity (FVC) in liter
Force Expiratory Flow 50 (FEV50) | longitudinal monitoring of assessments carried out as part of routine care during 5 yrs
  Force Expiratory Flow 50 (FEV50) in liter
Forced Expiratory Flow 25-75 (FEV25-75) | longitudinal monitoring of assessments carried out as part of routine care during 5 yrs
  Forced Expiratory Flow 25-75 (FEV25-75) in liter
Residual Volume (RV) | longitudinal monitoring of assessments carried out as part of routine care during 5 yrs
  Residual Volume (RV) in liter
Total Pulmonary Capacity | longitudinal monitoring of assessments carried out as part of routine care during 5 yrs
  Total Pulmonary Capacity in liter
Lung Clearance Index - Lung Clearance Index | longitudinal monitoring of assessments carried out as part of routine care during 5 yrs
  Lung clearance of nitrogen
colonization of bronchial secretions | longitudinal monitoring of assessments carried out as part of routine care during 5 yrs
  bacteria, fungi, mycobacteria
quality of life questionnaire | longitudinal monitoring of assessments carried out as part of routine care during 5 yrs
  CFQ questionnaire for children above 8 years: worse 0, better 100
ENT quality of life questionnaire | longitudinal monitoring of assessments carried out as part of routine care during 5 yrs
  SN-score: better score 1, worse 7
Abdominal quality of life questionnaire | longitudinal monitoring of assessments carried out as part of routine care during 5 yrs
  better score: 0, worse: 25
liver ultrasound | longitudinal monitoring of assessments carried out as part of routine care during 5 yrs
  liver ultrasound
elastometry (data available in centers with the necessary equipment) | longitudinal monitoring of assessments carried out as part of routine care during 5 yrs
  elastometry (data available in centers with the necessary equipment)
sweat test | longitudinal monitoring of assessments carried out as part of routine care during 5 yrs
  sweat collection
serum and fecal pancreatic biological markers | longitudinal monitoring of assessments carried out as part of routine care during 5 yrs
  immunoreactive trypsin, lipase, amylase, vitamin A and E, Prothrombin time, and fecal (fecal elastase
bone biological markers | longitudinal monitoring of assessments carried out as part of routine care during 5 yrs
  25OHvitD, Ca, P, PTH, Osteocalcin, IgF1, IgF1BP3, CTX
bone maturation | longitudinal monitoring of assessments carried out as part of routine care during 5 yrs
  Zscore (in relation to height and sex and weight) (data available in centers with the necessary equipment)
puberty | longitudinal monitoring of assessments carried out as part of routine care during 5 yrs
  serum dosage of FSH, LH, Estradiol, testosterone Pelvic ultrasound if puberty initiated in girls
intestine inflammation | longitudinal monitoring of assessments carried out as part of routine care during 5 yrs
  fecal Calprotectine
glycemic regulation | longitudinal monitoring of assessments carried out as part of routine care during 5 yrs
  monitoring of glycemic dysregulation ( as routinely done in the centers)
side effects: declarative collection and monitoring | longitudinal monitoring of assessments carried out as part of routine care during 5 yrs
  declarative collection and monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Sermet-Gaudelus, MD PhD, Principal Investigator — Société Francaise de la Mucoviscidose
Locations (1):
- Sermet-Gaudelus Isabelle, Paris, France

REFERENCES:
- [Derived] Sermet-Gaudelus I, Letierce A, Berteloot L, Bonnel AS, Chen Y, Makani P, Kelly-Aubert M, Kanoun F, Penalva L, Bouleghem N, Bihouee T, Bui S, Corvol H, Houdouin V, Mittaine M, Tatopoulos A, Weiss L, Wizla N, Kapel N, Bessou A, Tiddens HAWM, Caudri D, Reix P, Marguet C; MODUL-CF study group. Effect of elexacaftor-tezacaftor-ivacaftor on bronchial dilatations in adolescents with cystic fibrosis: a multicentre prospective observational study. Lancet Respir Med. 2026 Jan;14(1):38-48. doi: 10.1016/S2213-2600(25)00248-6. Epub 2025 Oct 22. PMID 41138737